CLINICAL TRIAL: NCT06812949
Title: Echocardiographic Right Ventricular Evaluation in Assessment of ARDS Lung Recruitment (ECHO-REVEAL)
Acronym: (ECHO-REVEAL)
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bari (Other)
Collaborators: Erasme University Hospital (Other); Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Salvatore Grasso, Full Professor and Head of Intensive Care Department, University of Bari
Other Study IDs: Prot.2026/CEL
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: ARDS
Keywords: Right ventricle; ARDS; Acute Respiratory Syndrome; Heart-lung interaction; Right Ventricular Strain; Recruitment manouvres; Mechanical Ventilation; PEEP; critical care ultrasounds
MeSH Terms: interventions — Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High Recruitment-to-Inflation (R/I) Ratio Group: This cohort includes ARDS patients with a Recruitment-to-Inflation (R/I) ratio > 0.5, indicating high lung recruitability in response to increased PEEP. These participants undergo a structured PEEP titration protocol, where ventilatory and hemodynamic parameters are assessed at low PEEP (5 cmH₂O) and high PEEP (15 cmH₂O). The primary focus is on evaluating right ventricular function, pulmonary pressures, and systemic hemodynamics to determine if high recruitability is associated with better tolerance to PEEP without inducing RV dysfunction.
  Interventions: Diagnostic Test: PEEP Titration with Echocardiographic, Hemodynamic, and Ventilatory Measurements
- Low Recruitment-to-Inflation (R/I) Ratio Group: This cohort consists of ARDS patients with a Recruitment-to-Inflation (R/I) ratio < 0.5, signifying limited lung recruitability and an increased risk of lung overdistension when PEEP is raised. These participants undergo the same PEEP titration protocol, with echocardiographic and ventilatory assessments at 5 cmH₂O and 15 cmH₂O PEEP levels. The objective is to evaluate the hemodynamic impact of higher PEEP in patients with poor lung recruitability, particularly in terms of right ventricular strain, pulmonary vascular resistance, and systemic venous congestion.
  Interventions: Diagnostic Test: PEEP Titration with Echocardiographic, Hemodynamic, and Ventilatory Measurements

INTERVENTIONS:
Diagnostic Test: PEEP Titration with Echocardiographic, Hemodynamic, and Ventilatory Measurements — This intervention consists of clinical recruitment maneuvers performed in mechanically ventilated patients by adjusting positive end-expiratory pressure (PEEP) at two levels: low PEEP (5 cmH₂O) and high PEEP (15 cmH₂O). Throughout these maneuvers, echocardiographic imaging, hemodynamic assessments, and ventilatory measurements are performed to evaluate the cardiorespiratory effects of PEEP adjustments. Transthoracic echocardiography (TTE) is used to assess right ventricular function, pulmonary pressures, and venous congestion, while mechanical ventilator parameters are recorded to monitor lung mechanics and compliance.
  Other Names: Recruitment Maneuvers with Cardiorespiratory Monitoring

SUMMARY:
Study Goal The goal of this observational, multicenter study is to evaluate how positive end-expiratory pressure (PEEP) affects right ventricular (RV) function in patients with acute respiratory distress syndrome (ARDS) who are receiving mechanical ventilation. Researchers will assess the Recruitment-to-Inflation (R/I) ratio, a measurement used to determine whether increasing PEEP helps open the lungs or causes harmful effects on the heart and circulation.

Main Study Questions

This study aims to answer the following questions:

1. How does PEEP affect right heart function in ARDS patients?
2. Can the R/I ratio predict whether PEEP will have a beneficial or harmful impact on the heart?
3. Which echocardiographic parameters best detect changes in right ventricular function caused by PEEP?

Who Can Participate?

Patients will be included in the study if they meet the following criteria:

* Age: 18 to 80 years.
* Condition: Diagnosed with moderate-to-severe ARDS, with a PaO₂/FiO₂ ratio <200 mmHg (an indicator of severe breathing difficulty).
* Mechanical Ventilation: Receiving invasive ventilation with at least 5 cmH₂O of PEEP and in deep sedation (fully dependent on the ventilator).
* Cardiac Monitoring: Equipped with a MostCare Up or equivalent device for continuous heart function monitoring.
* Informed Consent: Given directly by the patient or through a legal representative.

Patients will not be included in the study if they:

* Have severe pulmonary hypertension (high pressure in the lungs, ≥70 mmHg).
* Have a tricuspid valve prosthesis or other implanted cardiac devices that interfere with echocardiographic imaging.
* Have undergone recent heart surgery (within the past month).
* Have severe tricuspid valve disease that makes it difficult to assess right heart function.
* Are hemodynamically unstable, requiring high doses of medication to maintain blood pressure.
* Have poor ultrasound imaging conditions that prevent accurate heart scans.
* Have recently had a pulmonary embolism or have known blockages in the pulmonary arteries.
* Are receiving extracorporeal membrane oxygenation (ECMO) support.

Study Procedures

Participants will undergo a series of tests to measure the impact of PEEP on lung and heart function:

1. Initial Airway Closure Test: Patients will be evaluated while on a low PEEP level of 5 cmH₂O for 10 minutes to confirm eligibility.
2. Recruitment-to-Inflation (R/I) Ratio Assessment:

   * PEEP will be adjusted between low (5 cmH₂O) and high (15 cmH₂O) levels.
   * Researchers will measure changes in lung mechanics and heart function using ultrasound.
3. Echocardiographic Heart Function Assessment:

   * Transthoracic echocardiography (TTE) will be performed at each PEEP level to assess the right ventricle (RV) and circulation in the lungs.
   * Researchers will measure RV strain, size, and blood flow to determine how the heart reacts to PEEP changes.
4. Data Collection:

oKey respiratory and hemodynamic parameters will be recorded, including heart strain, cardiac output, pulmonary artery pressure, and venous congestion.

Primary and Secondary Study Outcomes

* Primary Outcome: The study will evaluate how RV function changes in response to different PEEP levels, using 2D RV strain measurements as a key indicator.
* Secondary Outcomes: Researchers will assess:

  * How accurately echocardiographic measurements (e.g., TAPSE, FAC, VExUS score) detect changes in RV function.
  * The relationship between the VExUS score (a marker of venous congestion) and RV strain changes.
  * The sensitivity and specificity of echocardiographic findings in predicting heart function shifts under different PEEP levels.

Statistical Analysis

* Researchers will compare echocardiographic heart function results at high PEEP vs. low PEEP using statistical models.
* The relationship between the R/I ratio and RV function will be analyzed using correlation tests and logistic regression.
* Receiver Operating Characteristic (ROC) analysis will be used to determine which echocardiographic parameter best detects RV dysfunction when the R/I ratio is low.

Study Size and Impact The study aims to enroll 60 patients (30 per group) to ensure that results are reliable. This sample size was calculated to detect at least a 10% change in RV strain, with a 90% probability of identifying significant effects.

Expected Benefits of the Study This study will help critical care doctors better understand how to adjust PEEP settings to balance lung recruitment and heart function in ARDS patients. By identifying the best methods to detect right heart dysfunction early, this research could lead to improved ventilation strategies and better survival outcomes for patients with severe lung injury.m

ELIGIBILITY:
Inclusion Criteria:

* Patients within 1 week from the diagnosis of acute respiratory distress syndrome (ARDS), defined according to the Berlin criteria.
* Non-pregnant.
* Age greater than or equal to 18 years.
* Monitored through MostCare Up or any other system for cardiac output (CO) monitoring and with invasive CVP catheter.
* Able to provide written informed consent to participate in the study directly or by a delegate.

Exclusion Criteria:

* Patients with severe pulmonary hypertension for any causes, defined by am echocardiographic PAPs ≥ 70 mmHg.
* Patients with tricuspid valve prostheses or percutaneous implanted devices (Triclip).
* Patients recently (within 1 month) undergoing cardiac surgery involving pericardiotomy.
* Patients with pre-existing severe tricuspid regurgitation.
* Patients with haemodynamic instability requiring high-dose vasopressors and/or inotropic agents in which recruitment manoeuvre are not considered to be safe according to clinical judgement.
* Patients whose acoustic window does not allow for the acquisition of the measurements under examination with transthoracic echocardiography.
* Patients with documented moderate-to-severe pulmonary embolism or known pulmonary artery stenosis.
* Patients undergoing Extracorporeal Membrane Oxygenation (ECMO).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18-80 years) diagnosed with moderate-to-severe acute respiratory distress syndrome (ARDS) who are undergoing mechanical ventilation in intensive care units (ICUs) at participating medical centers. Participants will be recruited from tertiary care hospitals specializing in critical care and echocardiography, specifically from the Intensive Care Units (ICU) of the following institutions:
  1. Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari, Italy - Department of Intensive Care
  2. Hôpital Erasme, Université Libre de Bruxelles (ULB), Brussels, Belgium - Department of Intensive Care
  3. Centre Hospitalier Universitaire (CHU) Saint-Pierre, Brussels, Belgium - Department of Intensive Care The study focuses on critically ill patients requiring invasive mechanical ventilation, where PEEP titration and recruitment maneuvers are part of standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Association Between the Recruitment-to-Inflation (R/I) Ratio and Right Ventricular Dysfunction in Mechanically Ventilated ARDS Patients | Within 30 minutes of PEEP titration at both high and low PEEP levels.
  The primary outcome of this study is to determine whether an unfavorable Recruitment-to-Inflation (R/I) ratio (<0.5) is associated with right ventricular (RV) dysfunction in ARDS patients undergoing PEEP titration during mechanical ventilation. RV function will be assessed through 2D speckle-tracking echocardiography (STE) of the RV free wall longitudinal strain (RVFWS) at low PEEP (5 cmH₂O) and high PEEP (15 cmH₂O). The study hypothesizes that patients with an R/I ratio <0.5 will show a significant increase (less negative values) in RV strain at high PEEP, indicating impaired RV function due to excessive lung overdistension and increased pulmonary vascular resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Grasso, Medicine and Surgery, Study Chair — University of Bari Aldo Moro
Locations (3):
- Belgium (2):
  - Hôpital universitaire - CHU Saint-Pierre, Brussels, Brussels Capital
  - Hôpital Erasme - Cliniques universitaires de Bruxelles, Brussels, Brussels Capital
- Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations, patient confidentiality, and data protection regulations. The study involves sensitive clinical and echocardiographic data collected from critically ill patients in intensive care units, which are subject to strict privacy and institutional policies. Additionally, the study protocol does not include provisions for external data sharing. However, aggregated and anonymized results will be made available through scientific publications and conference presentations.

REFERENCES:
- [Background] Vieillard-Baron A, Schmitt JM, Augarde R, Fellahi JL, Prin S, Page B, Beauchet A, Jardin F. Acute cor pulmonale in acute respiratory distress syndrome submitted to protective ventilation: incidence, clinical implications, and prognosis. Crit Care Med. 2001 Aug;29(8):1551-5. doi: 10.1097/00003246-200108000-00009. PMID 11505125
- [Background] Zapol WM, Snider MT. Pulmonary hypertension in severe acute respiratory failure. N Engl J Med. 1977 Mar 3;296(9):476-80. doi: 10.1056/NEJM197703032960903. PMID 834225
- [Background] Vieillard-Baron A, Prin S, Chergui K, Dubourg O, Jardin F. Echo-Doppler demonstration of acute cor pulmonale at the bedside in the medical intensive care unit. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1310-9. doi: 10.1164/rccm.200202-146CC. No abstract available. PMID 12421740
- [Background] Banavasi H, Nguyen P, Osman H, Soubani AO. Management of ARDS - What Works and What Does Not. Am J Med Sci. 2021 Jul;362(1):13-23. doi: 10.1016/j.amjms.2020.12.019. Epub 2020 Dec 26. PMID 34090669
- [Background] WHITTENBERGER JL, McGREGOR M, BERGLUND E, BORST HG. Influence of state of inflation of the lung on pulmonary vascular resistance. J Appl Physiol. 1960 Sep;15:878-82. doi: 10.1152/jappl.1960.15.5.878. No abstract available. PMID 13784949
- [Background] Mahmood SS, Pinsky MR. Heart-lung interactions during mechanical ventilation: the basics. Ann Transl Med. 2018 Sep;6(18):349. doi: 10.21037/atm.2018.04.29. PMID 30370276
- [Background] Price LC, McAuley DF, Marino PS, Finney SJ, Griffiths MJ, Wort SJ. Pathophysiology of pulmonary hypertension in acute lung injury. Am J Physiol Lung Cell Mol Physiol. 2012 May 1;302(9):L803-15. doi: 10.1152/ajplung.00355.2011. Epub 2012 Jan 13. PMID 22246001
- [Background] Evrard B, Goudelin M, Giraudeau B, Francois B, Vignon P. Right ventricular failure is strongly associated with mortality in patients with moderate-to-severe COVID-19-related ARDS and appears related to respiratory worsening. Intensive Care Med. 2022 Jun;48(6):765-767. doi: 10.1007/s00134-022-06730-0. Epub 2022 May 12. No abstract available. PMID 35552780
- [Background] Repesse X, Charron C, Vieillard-Baron A. Acute cor pulmonale in ARDS: rationale for protecting the right ventricle. Chest. 2015 Jan;147(1):259-265. doi: 10.1378/chest.14-0877. PMID 25560864